CLINICAL TRIAL: NCT02905656
Title: Strategies to Promote Cessation in Smokers Who Are Not Ready To Quit (PACE)
Brief Title: Strategies to Promote Cessation in Smokers Who Are Not Ready To Quit
Acronym: PACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Tennessee (Other)
Responsible Party: Principal Investigator, Robert Klesges, Professor, Public Health Sciences, University of Virginia
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 15-04215-XP 0027114; 1R01CA193245-01A1 (NIH)
Record Dates: First submitted 2016-09-14; First posted 2016-09-19 (Estimated); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Smoking Cessation
Keywords: quitline; nicotine replacement therapy; tobacco intervention; smokers not ready to quit
MeSH Terms: conditions — Smoking Cessation | interventions — Crisis Intervention; Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | US Export: No

ARMS (4):
- Brief Advice (Placebo Comparator): Participants will receive brief advice to quit smoking, and be provided psycho-education citing health consequences and the positive impact on mortality and morbidity.
  Interventions: Behavioral: Brief Advice
- Motivational Interviewing (MI) (Experimental): Motivational interviewing (MI) is a collaborative conversation style for strengthening a person's own motivation and commitment to change. MI attempts to avoid a confrontational style and, instead, guides participants toward choosing to make a change in their behavior.
  Interventions: Behavioral: Motivational Interviewing
- Rate Reduction (RR) (Experimental): Participants will be informed of the strong medical evidence of systematic reductions in smoking behavior can lead to long-term smoking cessation. This condition will receive Nicotine Replacement Therapy in the form of gum.
  Interventions: Behavioral: Rate Reduction; Drug: Pharmacological
- MI + RR (Experimental): In this intervention, participants receive both the skills based rate reduction intervention and the more motivationally based MI intervention. This condition will receive Nicotine Replacement Therapy in the form of gum.
  Interventions: Drug: Pharmacological; Behavioral: MI+RR

INTERVENTIONS:
Behavioral: Brief Advice — Psychoeducation
  Arms: Brief Advice
Behavioral: Motivational Interviewing — Guides participants toward choosing to make a change in their behavior with a collaborative conversation.
  Arms: Motivational Interviewing (MI)
Behavioral: Rate Reduction — Reducing the number of cigarettes consumed.
  Arms: Rate Reduction (RR)
Drug: Pharmacological — Nicotine Replacement Therapy in the form of gum.
  Arms: MI + RR; Rate Reduction (RR)
Behavioral: MI+RR — Combination of reducing the number of cigarettes consumed while guiding the participant to make a change in their behavior.
  Arms: MI + RR

SUMMARY:
To our knowledge, no study has evaluated the independent effects of motivational interviewing and rate reduction, individually versus in combination, for motivating smokers who are not ready to quit (SNRTQ) to increase both quit attempts and tobacco abstinence. Given the disseminability and the fact that findings can be readily translated into the network of tobacco quitlines, we propose: (1) To test a tobacco quitline for SNRTQ, following methods that we have previously implemented and evaluated (HL-123978, CA-127964); (2) To randomize 828 SNRTQs to: (a) Brief Advice + typical smoking cessation resources (control group); (b) motivational interviewing format recommended by the Clinical Practice Guidelines; (c) behavioral and pharmacologic rate reduction, and (d) both motivational interviewing and behavioral and pharmacologic rate reduction. This design allows us to evaluate the independent and additive effects of motivational interviewing and rate reduction on quit attempts and smoking cessation.

We plan to evaluate the efficacy of the intervention utilizing point prevalence at the 12-month follow-up. The Society for Research in Nicotine and Tobacco consensus paper concluded that point prevalence (7 days without a cigarette, "not even a puff") is an appropriate measure in measuring long term outcome in cessation induction trials. Prolonged abstinence at the 12-month follow-up and quit attempts at the 2-, 4- and 6-month and the 12-month follow-up are secondary endpoints. Self-efficacy, level of smoking reduction, tobacco dependence, intentions, motivation, and confidence to quit, and intervention adherence (# sessions attended, amount of nicotine replacement therapy used) will be tested as important treatment mediators.

DETAILED DESCRIPTION:
On the Society for Research in Nicotine and Tobacco definition of a cessation induction trial, which is a treatment that promotes cessation among all smokers, including those not ready to quit.1 One implication of this design is that success is based on percent abstinent at a given point in time and do not tie a follow-up to a determined quit date (since smokers not ready to quit often don't typically set formal quit dates).

Investigators research led to a four condition treatment design as the main independent variable of interest. Participants will be randomly assigned to four treatment conditions: (1) Brief advice; (2) motivational interviewing; (3) rate reduction; and (4) combination of motivational interviewing and rate reduction. All four intervention conditions will receive three sessions once a week, ideally, but can extend to a 6 week time period, each approximately 30 minutes in length, provided over a period of 4 to 6 weeks, depending on the participant's circumstances. Upon the completion of the main components, Booster sessions will be administered in 2-month increments throughout the intervention period (2 month, 4 month, & 6 month follow-up) in conjunction with study assessments. The window for the Booster sessions will be as indicated above 2M, 4M, and 6M after enrollment, but we will continue to try and reach them to complete the booster session for 4 weeks. For example, 2 month booster window opens at 8 weeks after enrollment and we will try to complete that 2 month booster within 4 weeks. Twelve months after randomization, prolonged abstinence will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand English
* For the past 12 months, has smoked 5 or more cigarettes a day
* 18 years or older
* Planning on Quitting smoking someday
* Access to a telephone
* Willing and able to use NRT in the form of gum
* Not currently using chantix or wellbutrin

Exclusion Criteria:

* Planning to quit smoking cigarettes in the next 30 days
* Currently pregnant, breastfeeding, or planning to become pregnant in the next 12 months
* Currently using chantix or wellbutrin
* Diagnosed with an unstable heart condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 903 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2020-06-16 (Actual); Study Completion 2020-06-16 (Actual)

PRIMARY OUTCOMES:
Point Prevalence Tobacco Abstinence | 12 months from randomization
  Point prevalence (7 days without a cigarette, "not even a puff") is an appropriate measure in measuring long term outcome in cessation induction trials.

SECONDARY OUTCOMES:
Prolonged Tobacco Abstinence | 12 months from randomization
  Prolonged abstinence will be defined as continuous abstinence from the point of initial cessation (with a two week grace period around the cessation date).

CONTACTS AND LOCATIONS:
Overall Officials: Robert Klesges, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Tennessee Health Science Center, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Derefinko KJ, Bursac Z, Hand SB, Ebbert JO, Womack C, Klesges RC. Planning a Change Easily (PACE) for smokers who are not ready to quit: a telephone-based, randomized controlled trial. Addiction. 2022 Jun;117(6):1748-1757. doi: 10.1111/add.15796. Epub 2022 Feb 1. PMID 34985171

DOCUMENTS (1):
  • Informed Consent Form (2018-11-01): https://cdn.clinicaltrials.gov/large-docs/56/NCT02905656/ICF_000.pdf